CLINICAL TRIAL: NCT06861920
Title: Targeting Interindividual Variability in NSAID Responses to Mitigate Chronic Pelvic Pain Risk in Dysmenorrhea (NSAID HEAL)
Brief Title: NSAID Use for Treating Dysmenorrhea and Preventing Chronic Pelvic Pain (NSAID HEAL)
Acronym: NSAIDHEAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of Chicago (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Kevin Hellman, Senior Research Scientist (Endeavor Health), Research Associate Professor (University of Chicago), Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000081; R01HD116714 (NIH)
Record Dates: First submitted 2025-02-28; First posted 2025-03-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Dysmenorrhea; Chronic Pelvic Pain; Pelvic Pain
Keywords: Painful Periods; NSAIDs; Chronic Pelvic Pain; Pelvic Pain; Periods
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain | interventions — Naproxen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Drug Paradigm (Active Comparator): Participants in this arm will be given naproxen sodium (550mg) as the study treatment, along with extended release acetaminophen (650mg) as a rescue medication. Participants are instructed to take 1 dose of naproxen sodium every 12 hours during the first 48 hours of their menstrual period. If participants do not feel adequate pain relief within 2 hours of taking a dose of naproxen sodium, they can take 1 dose of acetaminophen; they can repeat this process again in another 2 hours if needed for pain relief. Participants are instructed to follow this regime during each menstrual period for 1-year. Participants will not know whether or not they have received naproxen sodium or placebo, but they will know that they have been give acetaminophen as an optional rescue medication.
  Interventions: Drug: Naproxen Sodium 550mg; Drug: Extended Release Acetaminophen (650 mg)
- Placebo Paradigm (Placebo Comparator): Participants in this arm will be given a placebo capsule that is visually identical to the active drug as the study treatment, along with extended release acetaminophen (650mg) as a rescue medication. Participants are instructed to take 1 dose of the placebo every 12 hours during the first 48 hours of their menstrual period. If participants do not feel adequate pain relief within 2 hours of taking a dose of the placebo, they can take 1 dose of acetaminophen; they can repeat this process again in another 2 hours if needed for pain relief. Participants are instructed to follow this regime during each menstrual period for 1-year. Participants will not know whether or not they have received naproxen sodium or placebo, but they will know that they have been give acetaminophen as an optional rescue medication.
  Interventions: Drug: Placebo; Drug: Extended Release Acetaminophen (650 mg)

INTERVENTIONS:
Drug: Naproxen Sodium 550mg — Participants will receive Naproxen Sodium 550 mg oral tablet, administered twice daily for the first 48 hours of their menstrual period, for 1-year. Naproxen Sodium is a nonsteroidal anti-inflammatory drug (NSAID) used for pain relief and inflammation reduction. 550 mg naproxen sodium is the highest FDA-approved starting dosage, equivalent to 500 mg naproxen; the sodium formulation quickens absorption.
  Other Names: Aleve
  Arms: Active Drug Paradigm
Drug: Placebo — Participants will receive a placebo oral tablet, identical in appearance to Drug X, administered twice daily for the first 48 hours of their menstrual period, for 1-year. The placebo contains inactive ingredients with no known therapeutic effect.
  Arms: Placebo Paradigm
Drug: Extended Release Acetaminophen (650 mg) — Participants may take extended release acetaminophen 650mg oral tablet as needed for breakthrough menstrual pain. Participants will be instructed to take 1 dose of acetaminophen after 2 hours of taking a dose of either naproxen sodium or placebo, only if needed for pain relief. They are able to take an additional dose of acetaminophen after 2 more hours have elapsed for continued breakthrough symptoms. Use of rescue medication will be monitored and recorded.
  Other Names: Tylenol

SUMMARY:
The goal of this clinical trial is to learn if NSAIDs (i.e. naproxen sodium) can treat menstrual pain and prevent the development of chronic pelvic pain in menstruating adults with painful periods. The main questions it aims to answer are:

* Can non-menstrual pelvic pain reduction be predicted by menstrual pain response to NSAIDs?
* Will participants with the largest reductions in multi-site sensitivity following NSAID therapy have the largest reductions in non-menstrual pelvic pain?

Researchers will compare naproxen sodium to a placebo (a look-alike substance that contains no drug) to see if naproxen sodium works to treat painful periods.

Participants will:

* Take naproxen sodium or placebo during several days of their menstrual period every month for 1 year.
* Complete computer questionnaires and tests from home every 3 months.
* Complete at-home urine tests to measure hormones every few days for 1-year.
* Use a pin-prick to collect a small spot of blood, and use a pad or tampon to collect a sample of menstrual blood, and bring it to the research site twice over a 1-year period.
* Come to the research site twice over a 1-year period to complete sensory assessments and undergo a blood draw.

The major goal of the study is to develop a multivariable statistical model (see https://grants.nih.gov/grants/guide/rfa-files/RFA-NS-24-021.html ) describing the factors that effectiveness of pain medication and risk for chronic pain

ELIGIBILITY:
Inclusion Criteria:

* aged 18-35
* individuals who menstruate, with painful periods
* regular menstrual cycles (every 22-35 days)

Exclusion Criteria:

* presence of active pelvic or abdominal malignancies (primary or metastatic)
* conditions associated with the absence of regular menses such as polycystic ovarian syndrome, pregnancy, or any current use of continuous hormonal medication or contraceptive
* unable to read or comprehend the informed consent in English
* presence of other diagnosed chronic back or pelvic pain conditions (including chronic back pain, fibromyalgia, bladder pain syndrome, irritable bowel syndrome, vulvar pain syndrome, and endometriosis-associated pelvic pain)
* having another diagnosed/symptomatic chronic pain condition besides migraines with an average pain score >3/10 in the last month when not consuming pain relievers, or that requires daily treatment with opioids (ex. hydrocodone, oxycodone, codeine, morphine, hydromorphone, tapentadol, tramadol) or neuromodulators (also known sometimes as antidepressants [ex. amitriptyline, nortriptyline, imipramine, duloxetine, milnacipran, venlafaxine] or antiseizure medications [ex. topiramate, gabapentin, pregabalin, carbamazepine, lamotrigine])
* current or past history of stomach ulcers
* current or past history of gastrointestinal (GI) bleeding
* diagnosis of peptic ulcer disease
* current or past history of renal disorders
* current or past history of adrenal dysfunction
* diagnosis of liver disorders
* diagnosis of chronic acid reflex (i.e. GERD)
* Diagnosis of Crohn's disease or ulcerative colitis
* Coagulopathy
* Prolactinoma
* Von Willebrand disease
* Platelet disorders
* High blood pressure that is difficult to manage
* gastrointestinal conditions or surgeries that affect naproxen absorption
* bleeding disorders
* heart failure
* a history of stroke
* a history of heart attack
* active genitourinary or sexually transmitted infection
* allergy to non-steroidal anti-inflammatory drugs (NSAIDs) or their ingredients
* individuals who take the following medications: anticoagulants (i.e. warfarin), lithium, diuretics, antacids, angiotensin-converting enzyme (ACE) inhibitors, methotrexate, cholestyramine, or probenecids.
* Unmanaged diabetes (i.e. Fasting Blood Glucose: ≥ 126 mg/dL (≥ 7.0 mmol/L), Non-Fasting/Random Blood Glucose: ≥ 200 mg/dL (≥ 11.1 mmol/L), Hemoglobin A1c (HbA1c): ≥ 6.5%)
* Uncontrolled thyroid function (i.e. Hypothyroidism (Underactive Thyroid): Thyroid-Stimulating Hormone (TSH): > 4.5 mIU/L (mild) or > 10 mIU/L (severe) Free T4: Below the lower end of the reference range (usually < 0.9 ng/dL)
* Hyperthyroidism (overactive thyroid) (i.e. TSH: < 0.4 mIU/L (Suppressed or undetectable), Free T4: Above the upper end of the reference range (usually > 2.0 ng/dL)
* Liver dysfunction (i.e. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or bilirubin (unless known diagnosis of Gilbert's syndrome) ≥ 1.5 times the upper limit of the reference range)
* Kidney dysfunction (i.e. Serum creatinine > 1.1 mg/dL.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
M1 = Non-Menstrual Pelvic Pain (NMPP) Mediation by Menstrual Pain | From enrollment to end of treatment at 1-year
  "Non-menstrual pelvic pain (NMPP) will be assessed as the average of bladder, bowel, and non-menstrual pelvic pain ratings (0-10 scale) on non-bleeding days, excluding the two days before menstruation. Daily menstrual pain will be recorded during Menses (0-10 scale). The primary outcome is the reduction in NMPP at cycles 3,6,9, and 12, modeled using structural equation modeling to examine mediation by menstrual pain response to NSAIDs, accounting for endometrial inflammation (effluent cytokine levels). The mediation effect (M1) will be quantified using standardized path coefficients and indirect effects with bootstrapped 95% confidence intervals to determine the proportion of the NSAID effect on NMPP reduction. This outcome ranges from -1 to +1, with positive values indicating a worsening and negative values indicating a better mediation outcome.
V1= Non-Menstrual Pelvic Pain (NMPP) mediation by Visceral-Visceral Convergence (VVC) | From enrollment to end of treatment at 1-year
  In a structural equation model, VVC (bladder pain at first urge on 0-100 visual analog scale) and Multimodal Hypersensitivity) (reflecting widespread increased experimental sensitivity during the visual task, audio task, pressure pain tests, cold pressor, and conditioned pain modulation) will be constructed as a latent variable) mediation of the effect of NSAIDS on reductions in NMPP using a structural equation model. The mediation effect (V1) will be quantified using standardized path coefficients and indirect effects with bootstrapped 95% confidence intervals to determine the proportion of the VVC effect on NMPP. This outcome ranges from -1 to +1, with positive values indicating an worsening outcome and negative values indicating a better outcome.
Change in Non-Menstrual Pelvic Pain (NMPP) adjusted for holistic factors | From enrollment to end of treatment at 1-year
  Non-menstrual pelvic pain (NMPP) will be measured as the average of bladder, bowel, and non-menstrual pelvic pain ratings (0-10 scale) on non-bleeding days, excluding the two days before menstruation. Change in NMPP over time will be modeled using Structural Equation Modeling, adjusting for uterine inflammation (effluent prostaglandin concentration), sex hormones (estradiol, progesterone), and psychosocial factors (anxiety, depression, stress, sleep). The change in NMPP will be reported on a -10 to +10 scale, where -10 indicates improvement and +10 indicates worsening.

OTHER OUTCOMES:
Trial effects of NSAIDs on Non-Menstrual Pelvic Pain (NMPP) | From enrollment to end of treatment at 1-year
  The impact of NSAIDs on non-menstrual pelvic pain (NMPP) will be assessed by comparing participants using NSAIDs to those on placebo. Treatment effects will be measured as the difference in NMPP scores between the NSAID and placebo groups over time (Baseline, 4, 8, and 12 months) using electronic daily diaries. NMPP will be recorded on a 0-10 scale, where 0 indicates no pain (better outcome) and 10 indicates severe pain (worse outcome)
Trial effects of NSAIDs on chronic pelvic pain | From enrollment to end of treatment at 1-year
  The impact of NSAIDs on chronic pelvic pain (CPP) will be assessed by comparing participants using NSAIDs to those on placebo. Treatment effects will be measured by the proportion of participants meeting diagnostic criteria for CPP based on electronic daily diaries at Baseline, 4, 8, and 12 months. CPP status will be reported as a percentage, where 0% indicates no CPP (best outcome) and 100% indicates all participants meeting CPP criteria (worst outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Endeavor Health, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share these HEAL common Data Elements (CDEs): 1. Pain Intensity (PEG), 2. PROMIS Pain Interference, 3. PROMIS Physical functioning/quality of life, 4. PROMIS Sleep, 5. Pain catastrophizing (Sullivan 1995), 6. PROMIS Depression, 7. PROMIS Anxiety, 8. Global Satisfaction with Treatment (PGIC), 9. Substance Abuse (TAPS 1). The investigators will also share these HEAL-recommended demographics: age, sex at birth, gender identity, ethnicity, race, highest level of education, employment status, relationship status, annual household income, applied for disability insurance, pain duration, and postal code. The investigators will also share several data elements that lack a unified standard.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Electronic copies of our research publications will be deposited in PubMed Central within four weeks of acceptance by a journal, complete with appropriate metadata to ensure discoverability and accessibility upon publication. All publications will be released under the Creative Commons Attribution 4.0 Generic License (CC BY 4.0) or an equivalent open-access license. There will be no embargo period for the public availability of our publications. The underlying primary data supporting our publications will be made widely accessible through DASH, a HEAL-compliant repository. To the extent feasible, The investigators aim to share the underlying primary data concurrently with the publication, ensuring immediate access. All primary data shared will be subject to the CC BY 4.0 license or an equivalent open-access license.
Access Criteria: The IPD will be widely accessible via DASH, a Heal-compliant registry.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Background] Tu FF, Datta A, Atashroo D, Senapati S, Roth G, Clauw DJ, Hellman KM. Clinical profile of comorbid dysmenorrhea and bladder sensitivity: a cross-sectional analysis. Am J Obstet Gynecol. 2020 Jun;222(6):594.e1-594.e11. doi: 10.1016/j.ajog.2019.12.010. Epub 2019 Dec 20. PMID 31870730
- [Background] Hellman KM, Roth GE, Dillane KE, Garrison EF, Oladosu FA, Clauw DJ, Tu FF. Dysmenorrhea subtypes exhibit differential quantitative sensory assessment profiles. Pain. 2020 Jun;161(6):1227-1236. doi: 10.1097/j.pain.0000000000001826. PMID 32168005
- [Background] Kmiecik MJ, Tu FF, Silton RL, Dillane KE, Roth GE, Harte SE, Hellman KM. Cortical Mechanisms of Visual Hypersensitivity in Women at Risk for Chronic Pelvic Pain. medRxiv [Preprint]. 2021 Jan 18:2020.12.03.20242032. doi: 10.1101/2020.12.03.20242032. PMID 33501463
- [Background] Shlobin AE, Tu FF, Sain CR, Kmiecik MJ, Kantarovich D, Singh L, Wang CE, Hellman KM. Bladder Pain Sensitivity Is a Potential Risk Factor for Irritable Bowel Syndrome. Dig Dis Sci. 2023 Jul;68(7):3092-3102. doi: 10.1007/s10620-023-07868-7. Epub 2023 Mar 7. PMID 36879177
- [Background] Kmiecik MJ, Tu FF, Clauw DJ, Hellman KM. Multimodal hypersensitivity derived from quantitative sensory testing predicts pelvic pain outcome: an observational cohort study. Pain. 2023 Sep 1;164(9):2070-2083. doi: 10.1097/j.pain.0000000000002909. Epub 2023 Apr 27. PMID 37226937
- See also: NSAID HEAL website — https://NsaidHeal.com
- See also: Lab Website — https://Cureperiodpain.org